CLINICAL TRIAL: NCT02654418
Title: A Randomized, Double-blind, Comparative, Effectiveness and Safety Study of SIC 8000 in Subjects Undergoing Endoscopic Mucosal Resection (EMR) of Colonic Lesions Equal to or Larger Than 2 cm
Brief Title: Safety Study of SIC 8000 in Subjects Undergoing Endoscopic Mucosal Resection (EMR) of Colonic Lesions Equal to or Larger Than 2 cm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmo Technologies Ltd (Industry)
Responsible Party: Sponsor
Organization: CosmoTech (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CB-17-04/01
Record Dates: First submitted 2016-01-07; First posted 2016-01-13 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-02

CONDITIONS: Adenomas
Keywords: colonic polyps ≥20 mm,; adenomas; polyps
MeSH Terms: conditions — Adenoma; Polyps

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SIC 8000, 10 mL ampoules (Experimental): Procedure/Surgery: Endoscopic Mucosal Resection of large colon polyps (greater than or equal to 20 mm in size) with SIC 8000 injectate solution.
  Interventions: Procedure: Endoscopic Mucosal Resection of large colon polyps (greater than or equal to 20 mm in size)
- reference comparator (Active Comparator): Procedure/Surgery: Endoscopic Mucosal Resection of large colon polyps (greater than or equal to 20 mm in size) with Reference Comparator Injectate solution (site standard of care injectate solution).
  Interventions: Procedure: Endoscopic Mucosal Resection of large colon polyps (greater than or equal to 20 mm in size)

INTERVENTIONS:
Procedure: Endoscopic Mucosal Resection of large colon polyps (greater than or equal to 20 mm in size)

SUMMARY:
SIC 8000 is indicated for use in gastrointestinal endoscopic procedures for submucosal lift of polyps, adenomas, early-stage cancers or other gastrointestinal mucosal lesions, prior to excision with a snare.

DETAILED DESCRIPTION:
SIC 8000 is indicated for use in gastrointestinal endoscopic procedures for submucosal lift of polyps, adenomas, early-stage cancers or other gastrointestinal mucosal lesions, prior to excision with a snare.

The current trial will focus on only colonic polyps ≥20 mm removed by snare EMR technique.

Patients with lesions not suitable for EMR because of features strongly suggestive of sub-mucosal invasion will not be included.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of treatment naïve, laterally spreading sessile, flat polyps or adenomas of the colon equal to or greater than 20 mm in largest dimension, assessed by the investigator to be suitable for EMR.
2. The base of the lesion should measure at least 20mm in at least one dimension.
3. A photograph demonstrating the lesion size ≥20 mm against a stiff Boston Scientific Captivator snare of 20 mm must be recorded for each patient prior to randomization.
4. ASA status: limited anesthesiology risk, with ASA score 1, 2 or 3.
5. Contraception: women of childbearing potential must use at least one reliable method of contraception or be abstinent. Women of non-child-bearing potential or in post-menopausal status must have been in that status for at least 1 year. For all women of child-bearing potential, serum pregnancy test result must be negative at screening.
6. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study.
7. Informed consent: signed written informed consent must be completed before inclusion in the study.

Exclusion Criteria:

1. Age: Subjects under 18 years old are excluded
2. Consent: Subjects who refuse or who are unable to consent, vulnerable subjects are excluded.
3. Pregnancy: Pregnant or breastfeeding women
4. ASA status: High anesthetic risk (ASA score > 3)
5. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
6. Study participation: Subjects currently enrolled in any other clinical study or previous enrollment in a clinical study in the last 30 days
7. Subjects with Lesions less than 20 mm in largest dimension
8. Subjects with Lesions involving the muscularis propria (T2 lesions) on other staging modalities such as endoscopic ultrasonography (EUS)
9. Subjects with ulcerated depressed lesions (Paris type III) or biopsy proven invasive carcinoma
10. Presence of other malignant disease locally advanced or with metastasis
11. Presence of other lesions of the digestive tract as active Inflammatory colonic conditions (inflammatory bowel disease , e.g ulcerative colitis, Crohn's disease)
12. Endoscopic appearance of invasive malignancy
13. Previous treatment of the lesion (radiotherapy, endoscopy, surgery, chemotherapy) is exclusionary. Previous cold biopsy of the target lesion is not an exclusion criteria.
14. Previous partial resection or attempted resection of the target lesion is exclusionary.
15. Allergy: ascertained or presumptive hypersensitivity to study products; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study.
16. known or suspected gastrointestinal obstruction or perforation, toxic megacolon, active diverticulitis.
17. inflammatory bowel disease e.g ulcerative colitis or Crohn's 's disease
18. Hemostasis disorders (eg Von Willebran disease, haemophilia or factor V Leiden thrombophilia), known clotting disorder (INR>1.5 that cannot be corrected).
19. Other medical condition that in the investigator's opinion would make the administration of the study IMD or procedures hazardous to the subject.
20. Medical treatments (i.e.: radiotherapy, surgical endoscopic treatments) before the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2016-02; Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Sydney Resection Quotient (size of polyp in mm divided by number of resection pieces). | At V2 day of Endoscopic Mucosal resection of polyp (Day 1)
Proportion of subjects with en bloc resection of all endoscopically visible lesion | At V2 day of endoscopy (Day 1)

SECONDARY OUTCOMES:
Effectiveness compared to the reference comparator in terms of injected volume to provide initial polyp lift | At V2 day of Endoscopic Mucosal Reseaction (Day 1)
Injected volume required to complete the procedure | At V2 day of Endoscopic Mucosal Reseaction (Day 1)
Number of re-injections required to complete the procedure | At V2 day of Endoscopic Mucosal Resection (Day 1)
Number of resection pieces | At V2 day of Endoscopic Mucosal Reseaction (Day 1)
Ease of use rated on 5-point scale | At V2 day of Endoscopic Mucosal Reseaction (Day 1)
Time to resect the lesion completely | At V2 day of Endoscopic Mucosal Reseaction (Day 1)
Number of single session complete removal of lesions | At V2 day of Endoscopic Mucosal Reseaction (day 1)
Need for additional treatment modalities (eg coagulation, ablation, avulsion) | At V2 day of Endoscopic Mucosal Reseaction (Day 1)
Pathology negative report for lateral and/or deep margins | At V2 day of Endoscopic Mucosal Reseaction (Day 1)
Number of deep resections containing muscularis propria | At V2 day of Endoscopic Mucosal Reseaction (Day 1)
Histologically positive or negative Free margin confirmed in en-bloc resections | At V2 day of Endoscopic Mucosal Reseaction (Day 1)
  Histologist will assess if removed lesions have a free margin or not.
Recurrent or residual neoplasia confirmed by repeat standard endoscopy and biopsy (if applicable) at the follow up visit | Day 60 follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Dr Douglas Rex, Principal Investigator — Co-ordinating Investigator
Locations (5):
- United States (3):
  - Mayo Clinic, Jacksonville, Florida
  - Indiana University Hospital, Indianapolis, Indiana
  - Kansas City VA Hospital, Kansas City, Missouri
- Humanitas Research Hospital & Humanitas University, Milan, Italy
- Queen Alexandra Hospital, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Repici A, Wallace M, Sharma P, Bhandari P, Lollo G, Maselli R, Hassan C, Rex DK. A novel submucosal injection solution for endoscopic resection of large colorectal lesions: a randomized, double-blind trial. Gastrointest Endosc. 2018 Sep;88(3):527-535.e5. doi: 10.1016/j.gie.2018.04.2363. Epub 2018 May 8. PMID 29750983